CLINICAL TRIAL: NCT05800730
Title: Westlake Precision Nutrition Study 2 : Diet Challenges for Glucose Metabolism
Brief Title: Westlake Precision Nutrition Study 2 (WePrecision2)
Acronym: WePrecision2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 20230306ZJS001
Record Dates: First submitted 2023-03-23; First posted 2023-04-06 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-03

CONDITIONS: Healthy; Overweight and Obesity
Keywords: Personalized Nutrition; N-of-1; fasting; glucose metabolism; hair growth
MeSH Terms: conditions — Overweight; Obesity; Fasting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- refined carbohydrate breakfast (Breakfast A) (Experimental): white bread (50g) + milk powder (25g)
  Interventions: Other: refined carbohydrate breakfast
- whole grain breakfast (Breakfast B) (Experimental): plain oats (35g) + milk powder (25g)
  Interventions: Other: whole grain breakfast
- Energy-restricted diet (Experimental)
  Interventions: Other: energy-restricted diet
- time-restricted diet (Experimental)
  Interventions: Other: time-restricted diet

INTERVENTIONS:
Other: refined carbohydrate breakfast — After wearing CGM on Day 1, participants will be provided with breakfast A once daily on Day 3, Day 4, Day 7, Day 8, Day 10, Day 12. Breakfast A contains white bread (50g) and milk powder (25g). Since lunch and dinner would serve as wash-out meals, participants will be free to choose food but provide a record of their diets.
  Other Names: Breakfast A
  Arms: refined carbohydrate breakfast (Breakfast A)
Other: whole grain breakfast — After wearing CGM on Day 1, participants will be provided with Breakfast B once daily on Day 5, Day 6, Day 9, Day 11. Breakfast B contains plain oats (35g) and milk powder (25g). Since lunch and dinner would serve as wash-out meals, participants will be free to choose food but provide a record of their diets.
  Other Names: Breakfast B
  Arms: whole grain breakfast (Breakfast B)
Other: energy-restricted diet — After completing the baseline data and biological sample collection, the ERD group volunteers underwent a 10-day dietary intervention from day 3 to day 12. During this period, a standard breakfast was provided to all volunteers daily by the research staff through the school cafeteria. The ERD group volunteers still had their lunch and dinner provided by the research staff through the school cafeteria to ensure their daily energy intake was controlled between 1200-1500 kcal.
  Other Names: ERD
  Arms: Energy-restricted diet
Other: time-restricted diet — After completing the baseline data and biological sample collection, the volunteers in the TRD group will undergo a 10-day dietary intervention from day 3 to day 12. The TRD group needs to adjust their breakfast eating time to after 10:00 am daily, and they are free to choose their own lunch and dinner according to their dietary habits but must finish their meals before 4:00 pm. During this time window, no other energy-providing foods should be consumed.
  Other Names: TRD
  Arms: time-restricted diet

SUMMARY:
This is a dietary intervention study, which aims to explore different diet challenges for glucose metabolism, including carbohydrates and fasting dietary pattern. Considering the glucose responses to the same food are largely heterogeneous among people, this study integrates the concepts of precision nutrition and N-of-1 design. The study also aims to discover the different impact of the time-restricted diet (TRD) and the energy-restricted diet (ERD) on host metabolic health and our hair growth.

DETAILED DESCRIPTION:
The project is mainly based on classic field trial study design to compare impacts of different fasting patterns on host metabolic health. Under the condition of controlled diet background, individual N-of-1 study design is also organically integrated to compare personalized responses for standard meal tests. Participants will be required to wear continuous glucose monitoring (CGM) for 14 days. The diet intervention will be carried out after wearing CGM on Day 1. Then, all participants will be divided into three groups: energy-restricted diet (ERD), 18:6 time-restricted diet (TRD), and normal diet (ND). During Day 3 to Day 12, ERD restricts daily total energy intake within 1200-1500 kcal without meal timing limits, while TRD restricts the daily feeding window from 10:00 to 16:00, without total energy intake restriction. ND will maintain volunteers' original eating habits and rhythms as the control group. Individual N-of-1 trial design will be employed to all participants during Day 3 to Day 12 to compare the difference of postprandial glucose response to white bread or plain oats. These two standard breakfasts will appear in pseudo-random order. The TRD group needs to adjust the breakfast time to after 10:00 in the intervention periods.

ELIGIBILITY:
Inclusion Criteria:

* Participants have completed WePrecision trial in 2021
* Participants reside in Hangzhou
* Participants have no traveling plans within 3 months

Exclusion Criteria:

* Participants with metabolic diseases including diabetes, hypertension and cardiovascular diseases (CVD)
* Participants with craniocerebral trauma, cancer, liver disease, kidney disease, or other critical illness, or history of operation or medication
* Participants with bulimia nervosa, post-traumatic stress disorder (PTSD), chronic anxiety and depression or other critical neuronal disorder or history of relevant medication
* Being or to be pregnant or lactating.
* Participants with history of alcohol or drug addiction, or smoke above 15 cigarettes per day
* Concurrently participating other clinical trials.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Blood glucose profiling | 14 days
  Real-time blood glucose fluctuations will be recorded by CGM.
Change of glucose tolerance before and after intermittent fasting | Day 2 and Day 13
  Oral glucose tolerance test will also be conducted.

OTHER OUTCOMES:
Changes of fecal and urine metabolomics profiling | Day 2 and Day 13
  Fecal and urine metabolite extracts will be analyzed by performing liquid
Changes of serum metabolomics profiling | Day 2 and Day 13
  Targeted metabolomics are analyzed based on serum.
Changes of interleukin-1β (IL-1β), IL-6, IL-12 | Day 2 and Day 13
  Serum inflammatory factors (including IL-1β, IL-6, and IL-12) will be tested by enzyme-linked immunosorbent assay (ELISA) in pg/mL.
Changes of tumor necrosis factor-α (TNF-α) | Day 2 and Day 13
  Serum level of TNF-α will be tested by ELISA in ng/ml.
Changes of serum dopamine | Day 2 and Day 13
  Dopamine will be analyzed by serum.
Changes of lipid metabolism | Day 2 and Day 13
  Triglyceride, cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol, apolipoprotein A1 and apolipoprotein B.
Changes of weight | Day 2 and Day 13
  Weight will be measured in kilograms.
Height | Day 2
  Height will be measured in centimeters.
Body composition | Day 2
  Body composition (fat mass, lean mass in kg ) are assessed by bioelectrical impedance analysis.
Changes of both systolic and diastolic blood pressure | Day 2 and Day 13
  Both systolic and diastolic blood pressure will be measured in mmHg.
Hair | Day 2 and Day 13
  Hair sample and the hair growth will be measured in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (1):
- Westlake University, Hangzhou, Zhejiang, China